CLINICAL TRIAL: NCT06836544
Title: Efficacy of the ALL YOU NEED is LOVE Healthcare Transition Syllabus Among Pre- and Posttransplant Adolescents in Cali, Colombia
Acronym: Transition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Clinica Valle del Lili (Other)
Collaborators: International Society of Nephrology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 118-2016
Record Dates: First submitted 2025-02-10; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-01

CONDITIONS: Renal Transplant
Keywords: Pediatric nephrology; Educational; Healthcare transition; Kidney failure
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- "ALL YOU NEED IS LOVE" syllabus (Spanish version) (Experimental): ALL YOU NEED IS LOVE syllabus in 6 weeks program
  Interventions: Behavioral: ALL YOU NEED IS LOVE syllabus

INTERVENTIONS:
Behavioral: ALL YOU NEED IS LOVE syllabus — 1. Week 1: Introduction to the Kidneys
  2. Week 2: Chronic Kidney Disease, Medication Management
  3. Week 3: Making Healthy Choices
  4. Week 4: Learning about Self-Care
  5. Week 5: Becoming Independent
  6. Week 6: Review and Self-assessment

SUMMARY:
Background: To achieve optimal outcomes, adolescents with chronic or end-stage kidney disease must undergo healthcare transition (HCT) preparation from a pediatric- to an adult-focused setting. The pediatric nephrology group at the Fundación Valle del Líli in Cali, Colombia, collaborated with the University of North Carolina Chapel Hill STARx Program and Hospital Infantil de México Federico Gómez to start an HCT preparation program using their tools. The objective of this study was to evaluate the efficacy of the "ALL YOU NEED IS LOVE" syllabus (Spanish version) and its effects on HCT readiness in young patients with kidney failure, including renal transplants.

Methods: A pre-test/post-test quasi-experimental study was conducted without control group in 11- to 21-year-old consecutive patients with kidney failure followed at the Fundación Valle de Lili. Using the TRxANSITION Index, HCT readiness skills were measured before and after implementing the "ALL YOU NEED IS LOVE" syllabus, an educational curriculum delivered in three monthly 2-hour sessions. Analysis was performed using linear mixed models in R Studio software to evaluate intervention effects while accounting for participant characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 11 to 21 years along with their primary caregivers
* Either renal transplant recipients or in a renal transplant protocol
* Under follow-up by the Nephrology Service at Fundación Valle del Lili.

Exclusion Criteria:

* Patients were excluded if they did not sign the informed consent and/or assent to participate in the study.
* If they lost their care agreement with Fundación Valle del Lili due to administrative reasons related to their health insurance provider

Ages: 11 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of the "ALL YOU NEED IS LOVE" syllabus | 1 year
  The STARx questionnaire (SELF-MANAGEMENT AND TRANSITION TO ADULTHOOD WITH RX=TREATMENT) contains three subdomains that focus on three different areas of transition related knowledge - communication with medical provider, disease knowledge, and self-management.
  Each item is scored individually and worth a maximum of 5 points. Each item is answered by the patient on a 1 - 5 Likert scale and receive a corresponding score of 1 - 5 points for each item. Subdomain scores are combined to create a total score, ranging from 0 - 90.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Betz CL, Ferris ME, Woodward JF, Okumura MJ, Jan S, Wood DL. The health care transition research consortium health care transition model: a framework for research and practice. J Pediatr Rehabil Med. 2014;7(1):3-15. doi: 10.3233/PRM-140277. PMID 24919934
- [Derived] Forero-Delgadillo JM, Ochoa Jimenez VA, Padilla-Guzman A, Santamaria-Suarez MDP, Gonzalez-Fernandez MC, Medeiros M, Parraga P, de Ferris MED, Barbosa MM, Portilla-Buenaventura AM, Restrepo JM. Efficacy of the ALL YOU NEED IS LOVE healthcare transition syllabus among pre- and posttransplant adolescents in Cali, Colombia. BMC Nephrol. 2025 Apr 15;26(1):192. doi: 10.1186/s12882-025-04092-5. PMID 40234817